CLINICAL TRIAL: NCT04142268
Title: Comparison of Longitudinal Blood Pressure and Arterial Stiffness in Preeclamptic and Normotensive Women After Delivery: One-Year Follow-Up Results
Brief Title: Comparison of Longitudinal Blood Pressure and Arterial Stiffness in Preeclamptic Women After Delivery
Status: Completed | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Collaborators: Seoul National University Bundang Hospital (Other)
Responsible Party: Principal Investigator, Jung-Won Suh, Principal investigator, Seoul National University Hospital
Other Study IDs: B-1402-240-006
Record Dates: First submitted 2019-10-22; First posted 2019-10-29 (Actual); Last update posted 2019-10-29 (Actual); Status verified 2019-10

CONDITIONS: Preeclampsia and Eclampsia; Stiffness, Aortic; Blood Pressure
Keywords: Preelampsia; Cardio-ankle vascular index (CAVI); Aortic stiffness; Blood pressure; LDL-cholesterol
MeSH Terms: conditions — Pre-Eclampsia; Eclampsia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Preeclampsia group: PE was defined as diastolic BP of at least 110 mmHg on one occasion or diastolic BP of at least 90 mmHg on two consecutive occasions more than 4 hours apart, in combination with proteinuria (≥300 mg total protein in a 24-hour urine collection and, if this was not available, ≥+2 proteinuria by dipstick analysis on two consecutive occasions at least 4 hours apart) that develops after 20 weeks of gestation in previously normotensive women
- Control group: Normal pregnancy group

SUMMARY:
The investigator measured the arterial stiffness using cardio-ankle vascular index (CAVI) test in patient with preeclampsia and normal pregnant women to evaluate the longitudinal change of CAVI and their predictors.

DETAILED DESCRIPTION:
This study was a case control study and included 37 women with preeclampsia (PE group) and 36 normotensive women (control group) who gave birth to child at Seoul National University Bundang Hospital.

Cario-ankle vasuclar index (CAVI) was measured at one day, six months and one year after delivery in both group.

The investigator also checked the body weight, blood pressure, lipid profile, serum creatinine, aspartate transaminase (AST) and alanine transaminase (ALT) simultaneously with CAVI.

The relationship between the presence of preelampsia and longitudinal changes of CAVI, blood pressure and metabolic indices were evaluated using generalized estimating equation (GEE) method.

ELIGIBILITY:
Inclusion Criteria:

1. Case group : Women who were diagnosed preeclampsia based on the criteria of the International Society for the Study of Hypertension in Pregnancy
2. Control group : Normotensive women who gave birth to child at Seoul National University Bundang Hospital.

Exclusion Criteria:

* Women who were hemodynamically compromised or had bleeding complication after delivery were excluded.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: This study included 37 women with preeclampsia (PE group) and 36 normotensive women (control group) who gave birth to child at Seoul National University Bundang Hospital from March 2013 to May 2016.
Sampling Method: Probability Sample
Enrollment: 73 (Actual)
Dates: Start 2013-03 (Actual); Primary Completion 2016-10 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
The differences in longitudinal change pattern of CAVI between preeclampsia and normal pregnant women. | The CAVI was measured at one day, six months and one year after delivery in both groups.
  The CAVI was analyzed with generalized estimating equation (GEE) method to evaluate the different change pattern of CAVI between two groups.

SECONDARY OUTCOMES:
Systolic blood pressure | one day, six months and one year after delivery
  automated blood pressure, mmHg
Diastolic blood pressure | one day, six months and one year after delivery
  automated blood pressure, mmHg
Body weight | one day, six months and one year after delivery
  kilograms
Waist/Hip ratio | one day, six months and one year after delivery
  Waist circumference in centimeter, Hip circumference in centimeter, Waist/Hip Circumference Ratio is the ratio of waist circumference divided by hip circumference
Lipid profiles (Total cholesterol, TG, LDL, HDL) | one day, six months and one year after delivery
  mg/dL (milligrams per deciliter)
AST(aspartate aminotransferase), ALT(alanine aminotransferase) | one day, six months and one year after delivery
  IU/L (International Units Per Litre)
Serum creatinine | one day, six months and one year after delivery
  mg/dL (milligrams per deciliter)

CONTACTS AND LOCATIONS:
Overall Officials: Jung-Won Suh, MD, PhD, Principal Investigator — Seoul National University Bundang Hospital
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea

REFERENCES:
- [Derived] Kim S, Lim HJ, Kim JR, Oh KJ, Hong JS, Suh JW. Longitudinal change in arterial stiffness after delivery in women with preeclampsia and normotension: a prospective cohort study. BMC Pregnancy Childbirth. 2020 Nov 11;20(1):685. doi: 10.1186/s12884-020-03374-0. PMID 33176736